CLINICAL TRIAL: NCT07036536
Title: The NEET Registry: a Prospective, Observational Study for Outcomes of Non-euploid Embryo Transfers (NEET)
Brief Title: Non-Euploid Embryo Transfer (NEET) Registry
Status: Recruiting | Type: Observational
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Collaborators: CooperSurgical Inc. (Industry); Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: INC-NR-2024-006
Record Dates: First submitted 2024-10-02; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Infertility; Mosaicism; Aneuploidy
Keywords: IVF; PGT-A; aneuploid; FET
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The NEET Registry is a registry to track and study the outcomes of non-euploid embryo transfers (NEET) in The Prelude Network

DETAILED DESCRIPTION:
Preimplantation Genetic Testing for Aneuploidy (PGT-A) is widely offered as an option for patients pursuing pregnancy through in vitro fertilization (IVF). Most often, embryos with normal chromosome results are selected for transfer, with well established outcomes. However, for patient specific reasons, transferring an embryo with a non-euploid result (i.e. mosaic, isolated segmental aneuploid or aneuploidy of whole chromosome(s)) may be considered. Very little information is available on the long-term outcomes of mosaic embryo transfer. Even less has been published on outcomes for other types of non-euploid results. This study aims to collect prenatal, neonatal and pediatric outcome information for embryos transferred with the various types of non-euploid PGT-A results to better inform providers and patients in their decision making regarding such transfers.

ELIGIBILITY:
Inclusion Criteria:

* Patient is planning a non-euploid embryo transfer (NEET) at a fertility clinic in The Prelude Network.
* Patient has signed informed consent to participate in the registry.

Exclusion Criteria:

* Not applicable

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients planning a non-euploid embryo transfer (NEET) at a fertility clinic in The Prelude Network.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Embryo Implantation | 5 years
  The frequency of positive pregnancy test (blood serum QHCG) 10-14 days post embryo transfer

OTHER OUTCOMES:
Rate of Ongoing Pregnancy | 5 years
  The frequency of fetal heart tone identified on ultrasound post embryo transfer around 10-12 weeks gestation
Rate of Live Birth | 5 years
  The frequency of live birth post embryo transfer
Rate of Spontaneous Abortion | 5 years
  The frequency of spontaneous abortion post embryo transfer
Pediatric Developmental Milestones | 5 years
  Surveys inquiring about pediatric developmental milestones, as defined by the Center for Disease Control (CDC), are administered to the parent when child is 2 months, 6 months, 1 year, 2 year and 5 years of age. Results will be summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- Inception Fertility Research Institute, Houston, Texas, United States